CLINICAL TRIAL: NCT06560060
Title: Is the Gut Microbiome Associated With Residual Β-Cell Function and DeVElopment of Complications in Individuals With Longstanding Type 1 Diabetes Mellitus (MARVEL)
Brief Title: Do People With Complications of Type 1 Diabetes Mellitus Have a Different Microbiome (MARVEL)
Acronym: MARVEL
Status: Not yet recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Diabeter Nederland BV (Other)
Responsible Party: Principal Investigator, Max Nieuwdorp, prof dr, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL85375.018.23
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Type 1 Diabetes
Keywords: Microbiome; Type 1 diabetes; Complications; Betacell function
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA plasma: Determine changes in (microbial) metabolite composition. Metabolites will be measured by Metabolon via liquid chromatography-mass spectrometry for metabolomics. Measuring Pro-insulin/glucagon via ELISA
  EDTA buffycoat's: Isolate DNA and perform Immunochip
  Heparine plasma: Look at clinical chemistry
  Serum: Look at proteins
  Citrate plasma: Coagulation testing
  Feces samples: DNA will be isolated and used for shotgun sequencing on an Illumina platform to determine the microbiota composition.
  PBMC's: DNA isolation and subsequent HLA-typing and/or epigenetic analyses.
  Urine sample: UCPCR measurement
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MARVEL: 5000 individuals with type 1 diabetes > 18 years of age
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There are no interventions. The only medical procedure is a blood draw

SUMMARY:
This study looks at whether people with type 1 diabetes have different gut bacteria. We also want to see if this is linked to keeping insulin production up and preventing complications like heart disease and nerve damage. The aim is to find ways to keep more of the functions working, avoid low blood sugar and reduce diabetes complications.

DETAILED DESCRIPTION:
Rationale: It has become apparent that most individuals with type 1 diabetes mellitus (T1D) have some remaining β-cell function. Individuals with T1D and a preserved β-cell function have a lower risk of hypoglycemia and diabetic complications. The factors regulating residual β-cell function are unknown. A likely mechanism leading to β-cell preservation is regulation of immunological tone by the gut microbiome. Recently we published in a small pilot cohort (GUTDM1, METC 2020_105) that residual β-cell function is linked to better glycemic control (time in range) and linked to specific gut microbiota composition. Since this cohort was too small to also show a link with presence of diabetic complications and recruit enough individuals with preserved β-cell function for confirmatory intervention trials to increase β-cell function, we will now aim to recruit a larger follow-up cohort. The aim of this cohort is to a) investigate whether residual β-cell function is associated with gut microbiome composition and circulating immune cell counts in individuals with T1D and diabetic complications b) identify 500 potential eligible individuals with preserved β-cell function for future intervention trials.

Objective:

1. To investigate whether T1D individuals with preserved β-cell function exhibit a distinct gut microbial and circulating immune cell signature, leading to a reduced incidence of diabetes complications (CVD, nephropathy, neuropathy, and retinopathy).
2. Identify individuals with preserved β-cell function for diagnostics as well as future intervention studies to increase β-cell function.

Study design: 10-year longitudinal observational multicenter cohort study

Study population: 5000 individuals with type 1 diabetes >18 years of age, visiting the outpatient clinic of Diabeter center Amsterdam and Diabeter Nederland.

Main study parameters/endpoints: The primary endpoint is long-term residual β-cell function as assessed by baseline and stimulated 2-hour post meal urinary C-peptide levels at 3,6 and 10 years follow-up. The secondary endpoint pertains presence and incidence of diabetes complications (cardiovascular disease, nephropathy, neuropathy and retinopathy), gut microbiota composition measured in feces with shotgun sequencing, glucose time-in-range (CGM-metrics) and subsequent exogenous insulin dose. Tertiary endpoints include the profiling of immune cell subsets, assessment of autoreactive T lymphocytes and HLA typing by high resolution sequencing of circulating leukocytes (IMMOCHIP) in relation to untargeted plasma metabolomics (Metabolon).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: This study is considered a negligible-risk study. The patient will complete several questionnaires, keep track of a food diary and collect urine and feces prior to the baseline study visit. At the study visit we will require a fasted plasma sample, this will slightly increase the chances of a hypoglycemic episode, largely mitigated because all participants carry a continues glucose monitor. Additionally, we will calculate BMI, waist circumference, liver stiffness and measure blood pressure. The questionnaires inquire about the burden of diabetic complications, socio-economic status and financial literacy, abdominal complaints and hypoglycemic episodes, and comorbidities associated with diabetes, quality of life and psychological functioning. We argue that the risk and discomfort associated with this study is similar to the yearly diabetes check-up and justified in light of the potentially profound insights and novel treatments to be gained by studying the impact of the gut microbiome on residual β-cell function in T1D.

ELIGIBILITY:
Inclusion Criteria:

* All individuals with T1D visiting the outpatient clinic of Diabeter Center Amsterdam or Diabeter Nederland are potentially eligible if they are >18 years old.
* T1D diagnosis is made by the primary clinician prior to the study visit. Presence of auto- antibodies at time of diagnosis will be recorded.

Exclusion Criteria:

* Active infection during the study visit
* Inability or unwillingness to donate feces or urine.
* Smoking or illicit drug use (e.g. MDMA/amphetamine/cocaine/heroin/GHB) in the past three months or use during the study period.
* Inability or unwillingness to provide informed consent.
* Absence of a large bowel (ie colostomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population are patients with T1D in the Amsterdam region visiting the Diabeter Center Amsterdam which takes care for around +/- 5000 individuals with T1D.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2043-10-01 (Estimated); Study Completion 2043-10 (Estimated)

PRIMARY OUTCOMES:
Residual β-cell insulin secretion capacity: | At 0,3,6 and 10 years follow-up.
  assessed by non-invasive 2-hour post meal c-peptide release (residual β-cell function) in urine, composed of a urinary c-peptide to creatinine ratio (UCPCR).

SECONDARY OUTCOMES:
Presence and incidence of diabetes complications | At 0, 3, 6 and 10 years follow up
  cardiovascular disease, nephropathy, neuropathy, retinopathy and liver stiffness collected through medical history, yearly check-ups, bioimpadance measurement and questionnaires
Glycemic control: | At 0,3,6 and 10 years follow-up.
  changes in plasma biochemistry (glucose, HbA1c), glucose time in range (Freestyle Libre), urine (microalbuminuria) and subsequent exogenous insulin dose.
Intestinal microbiota composition | At 0,3,6 and 10 years follow-up.
  changes in gut microbiota composition as measured with shotgun sequencing in feces. Bristol stool chart for fecal composition.

OTHER OUTCOMES:
Circulating microbiota-derived metabolites | At 0,3,6 and 10 years follow-up.
  Changes in untargeted plasma metabolites.
Autoimmunity markers | At 0,3,6 and 10 years follow-up.
  HLA and immunotyping will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Henk-Jan Aanstoot, Dr., Principal Investigator — Diabeter Center Amsterdam/Diabeter Nederland; Max Nieuwdorp, Prof. Dr., Principal Investigator — Dept of Vascular Medicine, Amsterdam UMC - AMC; Nordin Hanssen, Dr., Principal Investigator — Dept of Vascular Medicine, Amsterdam UMC - AMC

IPD SHARING:
Plan to Share IPD: No